CLINICAL TRIAL: NCT04402216
Title: Using Virtual Reality Simulation to Prepare Children Undergoing MRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Colorado (Other)
Responsible Party: Principal Investigator, Brianne Newman, Certified Child Life Specialist, Children's Hospital Colorado
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20-0098
Record Dates: First submitted 2020-03-26; First posted 2020-05-26 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Anxiety; Distress
Keywords: anxiety; distress; virtual reality; MRI; pediatrics; child life; certified child life specialist; VR; preparation
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Current standard of care, no formal preparation (No Intervention): Participants in this group will receive the standard of care with no formal preparation. MRI technologist will meet patient prior to scan introducing role of patient, role of MRI technician, and give verbal discussion of MRI process. MRI technologist will offer opportunity for patient to watch a movie as alternative focus/distraction during MRI scan. The child life specialist will not meet with the caregiver or child during their visit.
- Child Life-led preparation (Experimental): Participants will meet with a child life specialist who will provide psychological preparation utilizing photos, MRI sounds, verbal discussion of MRI process, and discuss various coping strategies such as deep breathing or stress ball and option to watch a movie for alternative focus/distraction during the scan.
  Interventions: Behavioral: Child Life-led preparation
- MRI preparation video (Experimental): Participants will be shown an MRI preparation video by the research coordinator in the MRI dressing room prior to MRI scan. The MRI preparation video will walk the patient through the MRI experience with a mock patient explaining all the steps of MRI process from check in to discharge. The child life specialist will not meet with the caregiver or child during their visit.
  Interventions: Behavioral: MRI preparation video
- Child Life preparation with VR (Experimental): Participants will be provided MRI preparation with a child life specialist using the Kind VR device. The VR (virtual reality) session will consist of an audio and visual MRI experience designed to serve as an opportunity for the patient to practice their scan prior to MRI. The VR session will take place once during the Radiology admission and will be approximately 15 minutes in duration. The VR software was developed by Kind VR and was designed specifically for the purpose of preparation for brain MRI. The interactive VR experience walks patients through each step of an MRI. Patients can practice holding still for the MRI and will get feedback from the VR headset when they are moving their head. Along with VR practice session CCLS will discuss various coping strategies such as deep breathing and/or stress ball and option to watch a movie for alternative focus/distraction during the scan.
  Interventions: Behavioral: Child Life-led preparation; Behavioral: KindVR Virtual Reality MRI Preparation Experience

INTERVENTIONS:
Behavioral: Child Life-led preparation — Support from a certified child life specialist in preparation for MRI
  Arms: Child Life preparation with VR; Child Life-led preparation
Behavioral: MRI preparation video — A descriptive video about what to expect when undergoing MRI
  Arms: MRI preparation video
Behavioral: KindVR Virtual Reality MRI Preparation Experience — A VR experience to prepare pediatric patients for MRI, to be used in addition to support from a certified child life specialist
  Arms: Child Life preparation with VR

SUMMARY:
This study will evaluate the effectiveness of using virtual reality (VR) to reduce distress in pediatric patients undergoing MRI scans compared to other methods of preparation. Children will be divided into four groups. The investigators hypothesize the children who receive Child Life preparation with VR will experience decreased distress compared to the other 3 treatment groups (no formal preparation, Child Life-led preparation, and MRI preparation video). The investigators also hypothesize that children who receive Child Life-led preparation will experience better decreased distress than current standard of care (no formal preparation) and MRI preparation video.

DETAILED DESCRIPTION:
MRI scans can be difficult for children due to the confined space inside the MRI scanner, the loud noises that MRI scanners produce, and the amount of time that it takes to complete the scan. These factors can lead to a significant amount of distress and anxiety, both for the child undergoing the MRI scan and his or her family. Several techniques have been developed to reduce distress and anxiety in children undergoing MRI scans. Child Life Specialists have been proven to help reduce anxiety in children and better prepare them for MRI scans. Having a Child Life Specialist integrated into the multidisciplinary team treating a pediatric patient ensures that the child's emotional needs are being met as much as his or her physical needs.

Evaluation and intervention from a Child Life Specialist reduce anxiety and allows for children and families to be better prepared for their MRI, reducing distress of the child undergoing MRI, and reducing the need for anesthesia. Child life specialists are also able to utilize medical play using mock scanners and coach children in breathing exercises, such as blowing bubbles or pinwheels to help children comply with holding their breath during MRI scans, resulting in clearer images. Child Life specialists play a crucial role in effective communication with families and the rest of the medical team during and after examination.

III. Preliminary Studies/Progress Report

Another technique that has reduced distress in children during MRI is MRI compatible video goggles, which allow children to watch videos during the MRI scan. Giving children something to focus on while inside the MRI machine helps them to stay still and feel less anxious while still remaining awake. VR is a promising technology that has been used to reduce anxiety and serve as a pain distraction during intravenous placement required for MRI and CT scans as well as with children with sickle cell disease managing vaso-occlusive pain episodes. The inherent immersive and interactive properties of VR games make them effective for pain relief and distraction and also lends VR to countless potential applications in pediatric healthcare. KindVR is an independent VR firm that develops VR software specifically for the use of pediatric patients in a hospital setting. This software has been developed to minimize significant motion, mitigating risk of motion sickness or nausea, and providing targeted, age-appropriate content. There is not yet any published evidence that VR can be used to successfully prepare children for MRI scans, but there is strong evidence that this technology, especially paired with software specifically designed for use with pediatric patients in a hospital setting can impact important outcomes.

ELIGIBILITY:
Inclusion Criteria:

* (1) patients aged 6- 7 years who are scheduled for an MRI scan of the brain, face, orbitals, neck, spine, lower extremity, hip, humerus, knee, tibia and fibula, ankle, shoulder, elbow, forearm, hand, and/or wrist.
* (2) without anesthesia and
* (3) without contrast

Exclusion Criteria:

* (1) cognitive impairment that negates the use of the outcome tools or use of virtual reality device;
* (2) visual impairment that could not be corrected by lenses;
* (3) non-English speaking parent or patient.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 165 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Anxiety Rating | immediately before MRI scan
  Pre-procedural anxiety level of the child will be collected via child self-report and staff report before the MRI scan. Patient and Staff will report child's anxiety using a Visual Analog Scale with anchors "Not Anxious" and "Very Anxious." VAS scores will range from 1-100, with lower scores indicating less anxiety.

SECONDARY OUTCOMES:
Visit Satisfaction | immediately after MRI scan
  The caregiver will be given a standard Likert scale survey that rates satisfaction in the following areas: overall satisfaction with hospital visit, pain management, respect, and compassion. Guardians will be asked to select between "Very Satisfied," "Satisfied," "Neutral," and "Dissatisfied" in each of the aforementioned areas. The survey will also ask parents to rate teamwork between healthcare professionals and overall quality of care received by selecting a response of "Excellent," "Fair," "Neutral," and "Poor."
Demographic Information | collected retrospectively within 24 hours after verbal consent is obtained
  age, ethnicity, gender, type of MRI will be pulled via the electronic medical record retrospectively
MRI Scan Quality | immediately after MRI scan
  The MRI Technician will report whether the scan was complete, readable, and if rescanning was needed. Length of the MRI in minutes will be recorded as part of a procedural efficiency measure.
Technician feedback | immediately after MRI scan
  A cooperation rating will be collected from the MRI technician after the MRI scan. The technician will report the child's cooperation level using a Visual Analog Scale with anchors of "very uncooperative" and "very cooperative." VAS scores will range from 1-100, with lower scores indicating less cooperation.
Anxiety Rating | immediately after MRI scan
  Post-procedural anxiety level of the child will be collected via child self-report and staff report after the MRI scan. Patient and Staff will report child's anxiety using a Visual Analog Scale with anchors "Not Anxious" and "Very Anxious." VAS scores will range from 1-100, with lower scores indicating less anxiety.
Modified Yale Preoperative Anxiety Scale (m-YPAS) Distress Rating | collected while patient is MRI scan
  This structured, observational measure of preoperative anxiety in children consists of 27 items in five domains of behavior (Activity, Emotional Expressivity, State of arousal, Vocalization, and Use of parents). Using Kappa statistics, all m-YPAS domains have good to excellent inter- and intraobserver reliability; when compared with other global behavioral measures of anxiety, the m-YPAS had good validity.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
IDP will not be shared with other researchers.